CLINICAL TRIAL: NCT06659588
Title: Study of Populations at Risk of Developing Chronic Hepatitis Linked to Chronic Enteric Virus Infection in Patients With Primary Immunodeficiency and Secondary Humoral Deficiency
Acronym: EVAH
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231054; 2022-A02615-38 (Other: IDRCB Number)
Record Dates: First submitted 2024-02-15; First posted 2024-10-26 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Humoral Primary Immunodeficiencies (PIDs); Secondary Form of Humoral Immunodeficiencies; Combined Immunodeficiency (CID); Severe Combined Immunodeficiency (SCID)
Keywords: Humoral primary immunodeficiencies (PIDs); Secondary form of humoral immunodeficiencies; Combined immunodeficiency (CID); Severe combined immunodeficiency (SCID); Nodular regenerative hyperplasia; Chronic enteropathy; Enteric virus associated hepatitis
MeSH Terms: conditions — Severe Combined Immunodeficiency; Inflammatory Bowel Diseases | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Feces Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Humoral primary immunodeficiencies (PIDs): Patients with no age limit followed in one of the skills centers of the Reference Center for Hereditary Immune Deficits (CEREDIH) within the APHP (Necker-Enfants Malades Hospital, Saint-Louis Hospital and Cochin Hospital) for humoral primary immunodeficiencies.
  Interventions: Other: Plasma, urine and stool collection
- Secondary form of humoral immunodeficiencies: Patients with no age limit, followed in one of the skills centers of the Reference Center for Hereditary Immune Deficits (CEREDIH) within the APHP (Necker-Enfants Malades Hospital, Saint-Louis Hospital and Cochin Hospital) for a secondary form of humoral immunodeficiencies post anti-CD20 monoclonal antibody or post CAR-T cells therapy with alymphocytosis B and/or hypo IgA or IgM or IgG).
  Interventions: Other: Plasma, urine and stool collection
- Combined immunodeficiency (CID): Patients with no age limit followed in one of the skills centers of the Reference Center for Hereditary Immune Deficits (CEREDIH) within the APHP (Necker-Enfants Malades Hospital, Saint-Louis Hospital and Cochin Hospital) for a combined immunodeficiency.
  Interventions: Other: Plasma, urine and stool collection
- Severe combined immunodeficiency (SCID): Patients with no age limit followed in one of the skills centers of the Reference Center for Hereditary Immune Deficits (CEREDIH) within the APHP (Necker-Enfants Malades Hospital, Saint-Louis Hospital and Cochin Hospital) for a severe combined immunodeficiency beyond 2 years post cell therapy (allogeneic haematopoietic stem cell transplantation (aHSCT) or gene therapy).
  Interventions: Other: Plasma, urine and stool collection

INTERVENTIONS:
Other: Plasma, urine and stool collection — During a consultation for follow-up, we will take an extra-volume during a blood sample taken as part of the care. We will also collect stool and urine.
  There will be no biological collection for these samples. Organ biopsies carried out as part of the care (liver, kidney, digestive tract, spleen, lymph node) will also be studied as part of this research.

SUMMARY:
Dysimmune and specially hepatic immuno-pathological processes are frequent in patients with PIDs (primary immune deficiencies), particularly but not exclusively in patients with humoral defects. In the latter, nodular regenerative hyperplasia is a frequent complication. It is often associated with mislabeled chronic enteropathy. The investigators hypothesized that chronic viral infection with an enteric virus and the immune response that it implies might explain these processes.

To identify populations at risk of EVAH (enteric virus-associated hepatitis), four cohorts of patients will be studied:

* Primary humoral immune deficiencies
* Secondary humoral immune deficiencies (following anti-CD20 monoclonal antibodies, CAR-T cells)
* Combined immunodeficiencies
* Severe combined immunodeficiency syndrome (SCID) after allograft with humoral defect The investigators will collect clinical, biological and genetic information and features related to immunological responses and inflammatory damage for these patients. The investigators will include EVAH suspected patients and control patients in each cohort.

The investigators will take additional blood, stool and urine samples during the same time as the samples taken for the care.

The investigators will carry out tests for enteric viruses screening on stool, urine and plasma. The investigators will perform the viral screening on organ biopsies taken as part of the care.

A subgroup of representative patients (EVAH+ and EVAH-) will benefit from ancillary studies to characterize the leukocyte populations in the circulating blood and the immune response for these processes. In EVAH patients, the investigators will study specific anti-viral cellular response.

DETAILED DESCRIPTION:
Dysimmune and specially hepatic immuno-pathological processes are frequent in patients with PIDs (primary immune deficiencies), particularly but not exclusively in patients with humoral defects. In the latter, nodular regenerative hyperplasia is a frequent complication. It is often associated with mislabeled chronic enteropathy. The investigators hypothesized that chronic viral infection with an enteric virus and the immune response that it implies might explain these processes.

To identify populations at risk of EVAH (enteric virus-associated hepatitis), four cohorts of patients will be studied:

* Primary humoral immune deficiencies
* Secondary humoral immune deficiencies (following anti-CD20 monoclonal antibodies, CAR-T cells)
* Combined immunodeficiencies
* Severe combined immunodeficiency syndrome (SCID) after allograft with humoral defect The investigators will collect clinical, biological and genetic information and features related to immunological responses and inflammatory damage for these patients. The investigators will include EVAH suspected patients and control patients in each cohort.

The investigators will take additional blood, stool and urine samples during the same time as the samples taken for the care.

The investigators will carry out tests for enteric viruses screening on stool, urine and plasma by multiplex RT-PCR (Norovirus GI, Norovirus GII, Rotavirus, Sapovirus, and Astrovirus) and by targeted PCR (Enterovirus, Adenovirus, Aichi virus, Parechovirus, Kobuvirus and Astrovirus MLB1) on plasma and urine. The investigators will perform the viral screening on organ biopsies (liver, kidney, digestive tract, spleen, lymph node) taken as part of the care by mNGS (Metagenomics Next Generation Sequencing).

A subgroup of representative patients (EVAH+ and EVAH-) will benefit from ancillary studies to characterize the leukocyte populations in the circulating blood and the immune response for these processes. In EVAH patients, the investigators will study specific anti-viral cellular response by specific pentamers and elispot (enzyme-linked immunospot).

ELIGIBILITY:
Inclusion Criteria:

- Information and non-opposition from the legal representatives of minor patients, the patients themselves and adult patients of the population of interest.

Population of interest:

Patients with no age limit followed in one of the skills centers of the Reference Center for Hereditary Immunodeficiencies (CEREDIH) within the APHP (Necker-Enfants Malades hospital, Saint-Louis Hospital and Cochin hospital) and presenting:

* Humoral primary immunodeficiencies (PIDs) defined according to the IUIS (International Union of Immunological Societies) criteria
* Secondary form of humoral immunodeficiencies (post anti-CD20 monoclonal antibody or post CAR-T cells therapy with alymphocytosis B and/or hypo IgA or IgM or IgG)
* Combined immunodeficiency (CID) defined according to the IUES criteria
* Severe combined immunodeficiency (SCID) beyond 2 years post cell therapy (allogeneic haematopoietic stem cell transplantation (aHSCT) or gene therapy)

Exclusion Criteria:

* Patients not belonging to one of the target populations
* Opposition of legal representatives of minor patients, patients themselves and adult patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with no age limit followed in one of the skills centers of the Reference Center for Hereditary Immune Deficits (CEREDIH) within the APHP (Necker-Enfants Malades Hospital, Saint-Louis Hospital and Cochin Hospital) for humoral primary immunodeficiencies (PIDs), secondary form of humoral immunodeficiencies, combined immunodeficiency (CID), severe combined immunodeficiency (SCID).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-10-10 (Estimated); Study Completion 2026-10-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with chronic hepatic and/or digestive abnormalities | Day 0
  Number of patients with :
  * Chronic hepatitis (> 6 months with an increase in aspartate-aminotransferase/alanine-aminotransferase transaminases and/or gamma-glutamyl-transpeptidase levels greater than 2 times the upper limit of normal) without an identified cause (negative hepatotropic autoantibodies test and absence of infection by hepatitis viruses A, B, C, E).
  * Or histologically proven nodular regenerative hyperplasia.
  * And/or chronic enteropathy of undetermined etiology.
Number of patients with an identified enteric virus | Day 0
  The number of patients with an enteric virus identified in stools, and/or urine, plasma, organ biopsies and the type of enteric virus identified.
Statistical association between chronic hepatic and/or digestive abnormalities and enteric virus infection | Day 0
  We will use the homogeneity test Chi-square to compare the distribution of enteric virus groups (EVAH and controls).

SECONDARY OUTCOMES:
Description of characteristics of primary immunodeficiency of patients presenting enteric virus associated hepatitis (EVAH) | Day 0
  Clinico-biological characterization of patients presenting enteric virus associated hepatitis (EVAH) based on characteristics of immunodeficiency .
  * Genetic mutation or previous immunosupressor treatment
  * Plasma concentration of immunoglobulin in g/L
  * Lymphocytes (total and subpopulation) count in number of cells/mm3
  * Serological responses to antigen or vaccination : positive or negative
  Patients will be clustered in 4 cohorts :
  * Humoral primary deficiency
  * Secondary form of humoral immunodeficiencies
  * Combined immunodeficiency
  * Severe combined immunodeficiency Prevalence of EVAH patients will be evaluated in each subgroup
Description of global impact of chronic viral infection | Day 0
  Global impact of chronic viral infection will be evaluated by a clinical score including :
  * Clinical state alteration by Lansky score
  * BMI in kg/m^2
  * weight loss in kg
  * height stagnation in cm
  * chronic diarrhoea in number of watery stool/day
  * chronic abdominal pain : present or absent
  * presence of fever : present or absent
  * presence of neurological abnormalities : present or absent, description
  * haematological biological parameters : blood cells counts
  * renal function : creatinine blood concentration in µmol/L, Urea blood concentration in mmol/L, ionic blood concentration in mmol/L
  * Protein blood concentration in g/L
  * Presence of portal hypertension : presence or absence
  * presence of hepato-pulmonary syndrome : presence or absence The parameter will be compared between EVAH+ and EVAH- patients.
Microbiological characterization of patients presenting enteric virus associated hepatitis (EVAH) | Day 0
  The parameters will be compared between EVAH+ and EVAH- patients.
  Rate of patients with :
  * enteric virus in stools : presence or absence
  * enteric virus in urine : presence or absence
  * enteric virus in plasma : presence or absence
  * enteric virus in organ biopsies : presence or absence
Anatomic-pathologic characterization of patients presenting enteric virus associated hepatitis (EVAH) | Day 0
  The parameters will be compared between EVAH+ and EVAH- patients. Rate of patient with histologically proven
  * nodular regenerative hyperplasia : presence or absence
  * liver infiltrating T cell lymphocytes : presence or absence
Descrition of immunological characterization of patients presenting enteric virus associated hepatitis (EVAH) | Day 0
  The percentage of CD3+CD8+HLA-DRhigh CD38high CD127low will be mesured. The parameter will be compared between EVAH+ and EVAH- patients.
Phenotypically characterize the cellular response in EVAH patients | Day 0
  Characterize the immunological process associated with EVAH syndrome.
  The parameter will be compared between different cohorts of patients:
  - Percent (%) of leukocytes subpopulation in circulating blood by CyTOF
Transcriptionally characterize the cellular response in EVAH patients | Day 0
  Characterize the immunological process associated with EVAH syndrome. For a subgroup of representative patients (EVAH+ and EVAH-) the circulating leukocyte populations will be studied using single-cell RNA sequencing (scRNASeq).
  Comparison between different cohorts of patients.
Specific anti-viral responses in patients presenting enteric virus associated hepatitis (EVAH) | Day 0
  Identification and characterization of specific anti-viral cellular responses by specific pentamers and elispot in EVAH patients.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Michel, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Bénédicte Neven, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker-Enfants Malades, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riller Q, Fourgeaud J, Bruneau J, De Ravin SS, Smith G, Fusaro M, Meriem S, Magerus A, Luka M, Abdessalem G, Lhermitte L, Jamet A, Six E, Magnani A, Castelle M, Levy R, Lecuit MM, Fournier B, Winter S, Semeraro M, Pinto G, Abid H, Mahlaoui N, Cheikh N, Florkin B, Frange P, Jeziorski E, Suarez F, Sarrot-Reynauld F, Nouar D, Debray D, Lacaille F, Picard C, Perot P, Regnault B, Da Rocha N, de Cevins C, Delage L, Perot BP, Vinit A, Carbone F, Brunaud C, Marchais M, Stolzenberg MC, Asnafi V, Molina T, Rieux-Laucat F, Notarangelo LD, Pittaluga S, Jais JP, Moshous D, Blanche S, Malech H, Eloit M, Cavazzana M, Fischer A, Menager MM, Neven B. Late-onset enteric virus infection associated with hepatitis (EVAH) in transplanted SCID patients. J Allergy Clin Immunol. 2023 Jun;151(6):1634-1645. doi: 10.1016/j.jaci.2022.12.822. Epub 2023 Jan 10. PMID 36638922
- [Background] Klocperk A, Friedmann D, Schlaak AE, Unger S, Parackova Z, Goldacker S, Sediva A, Bengsch B, Warnatz K. Distinct CD8 T Cell Populations with Differential Exhaustion Profiles Associate with Secondary Complications in Common Variable Immunodeficiency. J Clin Immunol. 2022 Aug;42(6):1254-1269. doi: 10.1007/s10875-022-01291-9. Epub 2022 May 19. PMID 35589883
- [Background] Strohmeier V, Andrieux G, Unger S, Pascual-Reguant A, Klocperk A, Seidl M, Marques OC, Eckert M, Grawe K, Shabani M, von Spee-Mayer C, Friedmann D, Harder I, Gutenberger S, Keller B, Proietti M, Bulashevska A, Grimbacher B, Provaznik J, Benes V, Goldacker S, Schell C, Hauser AE, Boerries M, Hasselblatt P, Warnatz K. Interferon-Driven Immune Dysregulation in Common Variable Immunodeficiency-Associated Villous Atrophy and Norovirus Infection. J Clin Immunol. 2023 Feb;43(2):371-390. doi: 10.1007/s10875-022-01379-2. Epub 2022 Oct 25. PMID 36282455
- [Background] Fourgeaud J, Lecuit MM, Perot P, Bruneau J, Regnault B, Da Rocha N, Bessaud M, Picard C, Jeziorski E, Fournier B, Levy R, Marcais A, Blanche S, Frange P, Fischer A, Cavazzana M, Ferroni A, Jamet A, Leruez-Ville M, Eloit M, Neven B. Chronic Aichi Virus Infection As a Cause of Long-Lasting Multiorgan Involvement in Patients With Primary Immune Deficiencies. Clin Infect Dis. 2023 Aug 22;77(4):620-628. doi: 10.1093/cid/ciad237. PMID 37078608